CLINICAL TRIAL: NCT04864327
Title: The Effectiveness of a Tobacco Cessation Intervention Program Among Patients With Diabetes at Penang Hospital: a Randomised Controlled Trial
Brief Title: Smoking Intervention Among Patients With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansaa A.Ibrahim (Other Government)
Responsible Party: Sponsor-Investigator, Kansaa A.Ibrahim, Principal Investigator, Ministry of Health, Malaysia
Organization: Ministry of Health, Malaysia (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 9538; NMRR114779538 (Other: Clinical Research Centre (CRC))
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Smoking Cessation; Diabete Mellitus
MeSH Terms: conditions — Smoking Cessation; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Usual care
- intervention (Other): 5 minutes brief smoking cessation advise
  Interventions: Behavioral: Brief smoking cessation advise

INTERVENTIONS:
Behavioral: Brief smoking cessation advise — The tobacco cessation protocol consisted of performing a routine assessment (asking) of cigarette use; providing advice on the importance of quitting; performing an assessment of the tobacco user's readiness to quit; assisting in setting a quit date; and making arrangements for follow-up visits. This protocol is popularly known as the 5A's strategy (The first 3A's should be delivered to all smokers regardless of their willingness to quit). Tobacco users were identified by staff nurses. Clinicians provided brief advice on quitting, and the researcher assessed the patient's dependence and readiness to quit. Patients who were not ready to quit were motivated to consider quitting, whereas those who were ready to quit were referred to practitioners who could assist them and follow them in the tobacco cessation clinic
  Arms: intervention

SUMMARY:
This study determined the prevalence of tobacco smoking among patients with diabetes and evaluated the impact of a diabetes-specific tobacco cessation intervention on tobacco cessation outcomes and on the glycaemic control, blood pressure, lipid profile, complications, comorbidities and number of cigarettes consumed per day among the patients.

DETAILED DESCRIPTION:
The intervention protocol

Study Design and Study Population

This study is a randomized controlled trial involving diabetic patients who smoke tobacco, attending the diabetes clinic at Penang General Hospital in Malaysia. The prevalence of smoking among patients with diabetes will be measured by reviewing the patient who visit the Endocrine department within three months. The minimum sample size needed for calculating the prevalence estimated by using the equation below:

(Lwanga, S. K. and Lemeshow, S., 1991; Daniel, W. W., 1999; Cochran, W., 1977) n=(z^2 p (1-p))/d^2

Where n = the sample size; Z = the statistic for the 95% level of confidence used in the power analyses, which was 1.96; p = the expected prevalence or the proportion used, which was 0.5; and d = the precision used, which was 0.05. The estimated minimum sample size for the prevalence is 348 patients. One thousand one hundred eighteen medical records reviewed to find out the prevalence of smoking among the diabetic patients at the diabetes department in Penang General Hospital. Among those 1118 diabetic patients there were 108 smoking diabetic patients, depending on that; the prevalence of smoking among patients with diabetes will be 9.66%.

The study's participants will be randomly assigned into one of two groups: diabetes-specific tobacco cessation counseling group (intervention group) and the usual physician counseling group who will stay with the routine way in diabetes care counseling at Penang general hospital (control group). Study participants in the two groups will fill-up a questionnaire form to measure their knowledge, attitude, and practice of their physicians on smoking as a part of diabetes care and as a risk factor for its deterioration and complications pre and post the intervention.

Endocrinologists and physicians at the diabetic clinic will be asked to fill-up another questionnaire form to evaluate their attitude and practice in smoking cessation counselling among patients with diabetes and their willingness to apply the smoking cessation counselling in their clinics. All participants will sign an informed consent form to approve their agreement in their participation in the study.

Intervention Smoking Cessation Program among the Diabetic Patients The protocol of smoking cessation consists of a routine assessment (asking) about cigarette use, advice on the importance of quitting, an assessment of tobacco user's readiness to quit, assistance to set a quit date, and arranging for follow-up visits (Fiore, M. C. et al., 2008). This protocol is popularly known as the 5A's strategy. Tobacco users will be identified by staff nurses, clinicians will provide a brief advice on quitting and the researcher will assess patient's dependence and readiness to quit. Patients who are not ready to quit will be motivated to consider doing so, whereas those who are ready to quit will be referred to practitioners who can assist and follow them up in the smoking cessation clinic (American Diabetes Association, 2004).

All participants will be asked about their willingness to participate in the study, read the patient information sheet, and sign the patient consent form to approve their agreement to participate. Those who are willing to participate will be randomly assigned to either the intervention group (put letter I sticker on their records) or control group (put letter C sticker on their records). The assessment of readiness to quit smoking and nicotine dependence at baseline and after 3 and 6 months from the baseline will be done by filling the Fagerstrőm test questionnaire (FTQ) and Richmond test questionnaire. Patients will be followed for 6 months which is the standard follow-up duration for reporting data from clinical trials (Fiore, M. C. et al., 2008). Smoking abstinence or quitting will be confirmed by measuring the CO level using breath CO analyser at baseline and at 3 and 6 months of the intervention. Patients' glycaemic control, blood pressure, lipid profile, BMI, complication and comorbidities; also any quitting attempt during the study period will be recorded at the baseline and after 3 and 6 months as well from the patient's medical records and patients themselves.

The study's intervention will be delivered by physicians (who provide diabetes care to the participants), nurses and the smoking cessation clinic. The physicians will be trained on how to advise the diabetic patients to stop smoking and supported by a booklet that can help them for the wording in their counselling adapted from the guidelines. The smoking cessation clinic will help patients who are ready to quit by setting a quitting date and arranging follow-up visits for them. The intervention will be in compliance with the Malaysian guideline for the treatment of tobacco use and dependence using the 5 A's protocol (Ask, Advice, Assess, Assist, and Arrange for follow-up).

Randomization

In this study we use the Stat Trek's Random Number Generator to produce the random table to randomise the study population into two groups (control and intervention). Assuming that control group number 1 and intervention group is number 2 and we allow duplicate the values in the table and by choosing the random starting point described previously in this section.

ELIGIBILITY:
Inclusion Criteria:

Have a diagnosis of diabetes mellitus.

* Currently smoking tobacco.
* Speak English and/or Malay.

Exclusion Criteria:

* Do not have diabetes mellitus.
* Do not smoke tobacco or ex-smokers. do not speak English or Malay

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-05-05 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2012-12-01 (Actual)

PRIMARY OUTCOMES:
quitting rate | 12 months
  stop smoking
HbA1c | 12 months
  glucose level

SECONDARY OUTCOMES:
TriGlycerides, Low Density Lipoprotien, High Density Lipoprotien | 12 MONTHS
  LIPID PROFILE
BP(systolic and diastolic blood pressure) | 12 MONTHS
  BLOOD PRESSURE

CONTACTS AND LOCATIONS:
Overall Officials: Khansaa Albaroodi, Principal Investigator — PhD clinical pharmacy
Locations (1):
- Khansaa Albaroodi, Karbala, Others, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ibrahim AKA, Syed Sulaiman SA, Awaisu A, Shafie AA. Impact of brief smoking cessation intervention on quitting rate and glycemic control in patients with diabetes: a randomized controlled trial. J Int Med Res. 2023 Oct;51(10):3000605231208598. doi: 10.1177/03000605231208598. PMID 37890143